CLINICAL TRIAL: NCT02791581
Title: Understanding and Predicting Breast Cancer Events After Treatment (UPBEAT)
Brief Title: Understanding and Predicting Breast Cancer Events After Treatment
Acronym: UPBEAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00045463; WF 97415 (Other: Sponsor); 1R01CA199167-01 (NIH); NCI-2017-00386 (Registry Identifier: NCI Trial Identifier); NCI-2017-00386 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-05-20; First posted 2016-06-07 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Fatigue; Cardiovascular Events
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Breast Cancer Patients (Experimental): Breast cancer patients receiving non-anthracycline or anthracycline chemotherapy Cardiac MRIs will be performed baseline, 3 months (for cancer patients only), and 24 months.
  Baseline: Collect innovative MRI measures of CV function (LV and aorta); measurements of submaximal (6-minute walk) and, on 45% of the cohort, maximal (peak VO2) exercise capacity; questionnaire data to assess fatigue and behavioral and psychosocial risk factors; and biomarkers.
  Measurements will be repeated at 3±1, 12±2 and 24±2 months after initiation of chemotherapy treatment.
  Interventions: Diagnostic Test: Cardiac MRI
- Non-Cancer Controls (Experimental): Non-Cancer Controls Cardiac MRIs will be performed baseline and 24 months. Baseline: Collect innovative MRI measures of CV function (LV and aorta); measurements of submaximal (6-minute walk) and, 45% of the cohort, maximal (peak VO2) exercise capacity; questionnaire data to assess fatigue and behavioral and psychosocial risk factors; and biomarkers.
  Measurements will be repeated at 3±1, 12±2 (after the completion of radiation) and 24±2 months after initiation of baseline activities.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Breast Cancer Patients Cardiac MRIs will be performed baseline, 3 months (for cancer patients only), and 24 months.
  Non-Cancer Controls Cardiac MRIs will be performed baseline and 24 months.

SUMMARY:
This study is being done to see if patients receiving chemotherapy for breast cancer affects the heart, the ability to exercise and fatigue when compared to patients who do not have cancer.

DETAILED DESCRIPTION:
840 women aged ≥18 years old scheduled to receive chemotherapy for Stage I-III breast cancer and a comparison population of 160 women without cancer (1,000 total). Equal numbers of women will be recruited aged < 52 vs. > 52. At baseline, innovative MRI measures of CV function (LV and aorta); measurements of submaximal (6-minute walk) and, on 45% of the cohort, maximal (peak VO2) exercise capacity; questionnaire data to assess fatigue and behavioral and psychosocial risk factors; and biomarkers will be collected.

Measurements will be repeated at 3±1, 12±2 and 24±2 months. This study will assess the relevance of pre-existing factors such as age, black/white race, hypertension, smoking (yes/no), diabetes, coronary artery disease, menopause status, CV medications, and physical activity on the study outcomes. Also, this study will assess dynamic change in modifiable CV risk factors (including BMI, blood pressure, serum lipids, serum glucose, physical activity, psychosocial factors, lifestyle behaviors), and the cancer treatment including chemotherapy, radiation therapy, immunotherapy, and surgery.

ELIGIBILITY:
Inclusion Criteria for Women with Stage I - III Breast Cancer:

* Stage I-III female breast cancer (including inflammatory and newly diagnosed or locally recurrent breast cancer) but not metastatic breast cancer being treated with curative intent
* > 18 years old
* Scheduled to receive chemotherapy and/or estrogen antagonist aromatase inhibitors (anastrozole [Arimidex], letrozole [Femara], exemestane [Aromasin]).
* Able to hold breath for 10 seconds
* ECOG performance status 0 -2
* Able to walk at least 2 blocks without chest pain, dyspnea, shortness of breath or fainting
* Able to exercise on a treadmill or stationary cycle
* Participants in other ongoing clinical trials are eligible for this study

Exclusion Criteria for Women with Stage I-III Breast Cancer:

* Those with ferromagnetic cerebral aneurysm clips or other intracranial metal; pacemakers, defibrillators, functioning neurostimulator devices or other implanted non-compatible MRI devices (patients with tissue expanders will not be excluded)
* If previously measured, known LVEF <50%
* Symptomatic claustrophobia
* Unable to provide informed consent
* At the beginning of the study, pregnant women and women who are breast-feeding will not be enrolled.
* Severe pulmonary hypertension
* Within the past 6 months:

  * Acute pulmonary embolus
  * Deep vein thrombosis
* Within the past month:

  * Heart attack
  * Unstable or stable angina (cardiac chest pain)
  * Left main coronary artery disease
  * Symptomatic heart failure
  * Uncontrolled hypertension (SBP > 180 mm Hg or DBP > 120 mm Hg)
  * Severe valvular heart disease
  * Uncontrolled metabolic disease (diabetes with fasting BS >300 mg/dl, thyrotoxicosis, myxedema)
  * Aortic aneurism (>45 mm diameter) or aortic dissection
  * Uncontrolled slow or fast heart rhythm causing symptoms or hemodynamic compromise
  * Hypertrophic obstructive cardiomyopathy
* Patient does not understand English

Inclusion Criteria for Women Free of Cancer for Comparison:

* Healthy female without known coronary artery disease > 18 years old
* Able to hold breath 10 seconds
* ECOG performance status = 0 or 1
* Able to walk at least 2 blocks without chest pain, dyspnea, shortness of breath or fainting
* Able to exercise on a treadmill or stationary cycle
* No personal history of cancer other than superficial skin cancers
* Has never received chemotherapy, radiation therapy, immunotherapy, or had breast cancer related surgery
* If previously measured, LVEF ≥ 50%

Exclusion Criteria for Women Free of Cancer for Comparison:

* Inflammatory conditions such as lupus or inflammatory bowel disease
* Overt coronary artery disease or heart failure
* Those with ferromagnetic cerebral aneurysm clips or other intracranial metal; pacemakers, defibrillators, functioning neurostimulator devices or other implanted non-compatible MRI devices
* Symptomatic claustrophobia
* Unable to provide informed consent
* At the beginning of the study, pregnant women or women who are breast feeding will not be enrolled.
* Severe pulmonary hypertension
* Within the past 6 months:

  * Acute pulmonary embolus
  * Deep vein thrombosis
* Within the past month:

  * Heart attack
  * Unstable or stable angina (cardiac chest pain)
  * Left main coronary artery disease
  * Symptomatic heart failure
  * Uncontrolled hypertension (SBP > 180 mm Hg or DBP > 120 mm Hg)
  * Severe valvular heart disease
  * Uncontrolled metabolic disease (diabetes with fasting BS >300 mg/dl, thyrotoxicosis, myxedema)
  * Aortic aneurism (>45 mm diameter) or aortic dissection
  * Uncontrolled slow or fast heart rhythm causing symptoms or hemodynamic compromise
  * Hypertrophic obstructive cardiomyopathy
* Patient does not understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2034-07-31 (Estimated); Study Completion 2034-07-31 (Estimated)

PRIMARY OUTCOMES:
FACT-Fatigue | Baseline
  Participants rate the degree to which each item applies in the past 7 days prior to Baseline using a 5-point scale. Scores range from 0-52, with higher scores indicating greater fatigue.
Change in FACT-Fatigue Results | Baseline and 3 months
  Participants rate the degree to which each item applies in the past 7 days using a 5-point scale. Scores range from 0-52, with higher scores indicating greater fatigue.
Change in FACT-Fatigue Results | Baseline, 3 months and 12 months
  Participants rate the degree to which each item applies in the past 7 days using a 5-point scale. Scores range from 0-52, with higher scores indicating greater fatigue.
Change in FACT-Fatigue Results | Baseline, 3 months, 12 months and 24 months
  Participants rate the degree to which each item applies in the past 7 days using a 5-point scale. Scores range from 0-52, with higher scores indicating greater fatigue.
Change in MRI Exam Results | Baseline, 3 months and 24 months
  The exam will measure left ventricular volumes, ejection fraction, myocardial strain/strain rate, mass, mapping, aortic pulse wave velocity and aortic wall thickness. The exam will take 10 - 15 minutes to complete.
Change in 6 Minute Walk Results | Baseline, 3 months, 12 months and 24 months
  The purpose of this test is to find out how far the participant can walk in 6 minutes.

SECONDARY OUTCOMES:
Cohen's 4-item Perceived Stress Scale (PSS) | Baseline, 3 months, 12 months, and 24 months
  A summed scale asking how often over the prior two weeks four aspects of stress were experienced (1=never to 5=very often)
  o weeks four aspects of stress were experienced (1=never to 5=very often)
Cook-Medley Hostility Scale | Baseline
  A 14-item scale used to assess the effect of hostility associated with cardiovascular risk factors.
  Minimum Score: 0 Maximum Score: 13 Higher values indicate greater hostility.
Changes in FACT-Fatigue Results | Baseline, 3 months, 12 months, and 24 months
  Participants rate the degree to which each item applies in the past 7 days using a 5-point scale. Scores range from 0-52, with higher scores indicating greater fatigue.
6 Minute Walk Results | Baseline, 3 months, 12 months and 24 months
  The purpose of this test is to find out how far the participant can walk in 6 minutes.
RAND MOS 36-item Short Form Health Survey (SF-36) | Baseline, 3 months, 12 months and 24 months
  SF-36 consists of 36 items measuring the following 8 domains: physical function, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional health problems, and mental health. These 8 domains also provide two summary scores.
Center for Epidemiological Studies Depression Scale (CESD-10) | Baseline, 3 months, 12 months and 24 months
  Screening questionnaire assessing depressive symptoms during the last week
Godin Leisure-Time Exercise Questionnaire (LTEQ) | Baseline, 3 months, 12 months and 24 months
  Main process measure of physical activity participation
PACE Adult Sedentary Behaviors Survey | Baseline, 3 months, 12 months and 24 months
  Assess sedentary lifestyle behaviors
PROMIS Short Form 8A Measure of Sleep Disturbance | Baseline, 3 months, 12 months and 24 months
  Assess time course and risk factors associated with sleep disturbance and fatigue
  Minimum Score: Raw: 8, T-score: 28.9 Maximum Score: Raw: 40, T-score: 76.5 Higher values represent greater sleep disturbance.
PROMIS Applied Cognitive Abilities Short Form 8A and Applied Cognition General Concerns Short Form 8A | Baseline, 3 months, 12 months and 24 months
  Measurement of different aspects of cognitive functioning.
  PROMIS Applied Cognitive Abilities Short Form 8A
  - Minimum Score: Raw: 8, T-score: 27.0 Maximum Score: Raw: 40, T-score: 64.8 Higher values represent better cognition.
  Applied Cognition General Concerns Short Form 8A
  - Minimum Score: Raw: 8, T-score: 23.3 Maximum Score: Raw: 40, T-score: 62.7 Higher values represent better cognition.
Walking Efficacy for Duration Scale | Baseline, 3 months, 12 months and 24 months
  Comprised of six items and will be included as a measure of exercise capacity
Chair Stands - Measures Leg Strength | Baseline, 3 months, 12 months and 24 months
  Participants will be first asked to stand from a sitting position without using their arms. If they can perform the task, they will then be asked to stand up and sit down five times as quickly as possible. The time to complete the task will be recorded.
Standing Balance Test | Baseline, 3 months, 12 months and 24 months
  Participants will be asked to maintain balance for up to 30 seconds in three positions characterized by a progressive narrowing of the base support.
Gait Speed Test | Baseline, 3 months, 12 months and 24 months
  Participants will be instructed to start at a marked walking course with toes touching the start line and when cued to start, will begin walking at their ususal speed. The time to walk from the starting line to the end of the 4-meter walk will be recorded.
Grip Strength | Baseline, 3 months, 12 months and 24 months
  Grip strength is assessed with an isometric handgrip dynamometer while the participant is sitting with the head facing straight ahead. The elbow should be bent at a 90 degree angle and the wrist should be at the mid-prone position.
Range of Motion | Baseline, 3 months, 12 months and 24 months
  Range of motion at the shoulder joint will be assessed with shoulder flexion and shoulder abduction with a goniometer.
KCCQ-12 Questionnaire | Baseline, 24 months
  Independently measures the patient's perception of their health status which includes heart failure symptoms (frequency and burden), physical and social limitations, and how their heart failure impacts their QOL within a 2-week recall period.

OTHER OUTCOMES:
B-type natriuretic peptide (BNP) | Baseline and 24 months
  Serum BNP as a predictor of exercise intolerance
Troponin - 1 | Baseline and 3 months
  Acquired to determine associations between troponin levels during therapy and the onset of cardiac and vascular dysfunction, exercise capacity, and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hundley, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (66):
- United States (66):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu

REFERENCES:
- [Derived] Mabudian L, Reding K, D'Agostino RB Jr, Heiston EM, Bellissimo MP, Olson K, Ntim WO, Klepin HD, Dressler EV, Moore T, Jordan JH, O'Connell NS, Ladd A, Weaver KE, Ky B, Wagner LI, Hackney MH, Lesser GJ, Hundley WG; UPBEAT Study Team. The relationship between body composition and left ventricular performance in women with breast, lymphoma, or sarcoma cancer. Cardiooncology. 2024 Jun 6;10(1):34. doi: 10.1186/s40959-024-00233-1. PMID 38845066
- [Derived] Garg R, D'Agostino RB Jr, O'Connell N, Lesser GJ, Salloum FN, Hines AL, Melendez GC, Jordan JH, Ky B, Wagner LI, Sutton AL, Bottinor W, Olson KC, Ladd AC, Hundley WG; UPBEAT Study Team. Hypertension Severity and Declines in Left Ventricular Ejection Fraction Among Women Receiving Adjuvant Chemotherapy for Breast Cancer (WF-97415 UPBEAT). Hypertension. 2024 Jun;81(6):1365-1373. doi: 10.1161/HYPERTENSIONAHA.123.21817. Epub 2024 Apr 18. PMID 38634292
- [Derived] Bellissimo MP, Canada JM, Jordan JH, Ladd AC, Reding KW, Moore TL, Ntim WO, Heiston EM, Brubaker P, Mihalko SL, D'Agostino R Jr, O'Connell N, Ky B, Wagner LI, Hackney MH, Weaver KE, Lesser GJ, Avis NE, Sutton AL, Lucas AR, Franco RL, Fuemmeler BF, Salloum FN, Hundley WG; UPBEAT Study Group. Physical Activity During Breast Cancer Therapy Associates With Preserved Exercise Capacity and Cardiac Function (WF97415). JACC CardioOncol. 2023 Mar 21;5(5):641-652. doi: 10.1016/j.jaccao.2022.12.011. eCollection 2023 Oct. PMID 37969655
- [Derived] Bellissimo MP, Canada JM, Jordan JH, Ladd AC, Heiston EM, Brubaker P, Mihalko SL, Reding K, D Agostino R, O Connell N, Hackney MH, Weaver KE, Lesser GJ, Avis NE, Hundley WG. Changes in Physical Activity, Functional Capacity, and Cardiac Function during Breast Cancer Therapy. Cancer Epidemiol Biomarkers Prev. 2022 Jul 1;31(7):1509. doi: 10.1158/1055-9965.EPI-22-0470. PMID 35775211